CLINICAL TRIAL: NCT00653926
Title: Local Infiltration Analgesia (LIA) With Ropivacaine, Ketorolac and Epinephrine Intra- and Postoperatively in Unicompartmental Knee Arthroplasty
Brief Title: Local Infiltration Analgesia Following Unicompartmental Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Professor Kjell Axelsson, Dept. of Anaestesiology, Örebro University, Örebro, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAK-mini
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Local infiltration analgesia; Knee arthroplasty; Postoperative pain management following unicompartmental knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Group A (Active) receives a multimodal injection intra- and postoperatively
  Interventions: Drug: ropivacaine, ketorelac and epinephrine
- P (Placebo Comparator): Group P (Placebo) receives no injection intraoperatively and a saline injection postoperatively
  Interventions: Drug: saline

INTERVENTIONS:
Drug: ropivacaine, ketorelac and epinephrine — In Group A, 200 mg ropivicaine, 30 mg ketorelac and 0.5 mg epinephrine (total volume 106 ml) are infiltrated by the surgeon into the soft tissues peri-articularly during the operation in the following way: Before inserting the components, 20-30 ml are injected into the posterior capsule and before closure of the wound the rest is injected into the capsule incision, the synovium, the ligament and the subcutaneous tissue After 21 postoperative hours in Group A, 150 mg ropivicaine, 30 mg ketorelac and 0.1 mg epinephrine, total volume 22 ml, are injected intraarticularly via the catheter.
  Arms: A
Drug: saline — In Group P (placebo) no injections were given intaoperatively. All patients had a tunnelled intra-articular multihole 20-G catheter placed at the end of the operation by the surgeon.After 21 postoperative hours 22 ml of saline was injected intraarticularly via the catheter.
  Arms: P

SUMMARY:
The primary aim of this study is to evaluate if intra- and postoperative administration of ropivacaine, ketorolac and epinephrine into the operating field would affect hospital stay. Secondary end-points are morphine consumption, pain intensity and side effects. In an attempt to assess the safety of this technique, knee function and patient satisfaction scores are assessed up to 6 months after surgery.

DETAILED DESCRIPTION:
Postoperative pain is often severe following knee arthroplasty. Recently, a local infiltration analgesia (LIA) technique was developed by Drs Kerr and Kohan in Sydney, Australia. With this LIA-technique, a long-acting local anesthetic (ropivacaine), a nonsteroidal anti-inflammatory drug (ketorolac), and epinephrine are infiltrated intraoperatively and via an intraarticular catheter postoperatively.

The primary aim of this study is to evaluate if intra- and postoperative administration of ropivacaine, ketorolac and epinephrine into the operating field would affect hospital stay. Secondary end-points were morphine consumption, pain intensity and side effects. In an attempt to assess the safety of this technique, knee function and patient satisfaction scores were assessed up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unicompartmental knee arthroplasty
* Aged 20-80 yrs.
* ASA physical status I-III and mobility indicating normal postoperative mobilization

Exclusion Criteria:

* Known allergy or intolerance to one of the study drugs
* Serious liver-, heart- or renal decease
* Rheumatoid arthritis
* Chronic pain or bleeding disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study was to evaluate if intra- and postoperative administration of ropivacaine, ketorolac and epinephrine into the operating field would affect hospital stay. | April, 2007

SECONDARY OUTCOMES:
Secondary end-points were morphine consumption, pain intensity and side effects. In an attempt to assess the safety of this technique, knee function and patient satisfaction scores were assessed up to 6 months after surgery. | September, 2007

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Axelsson, Prof., Principal Investigator — Orebro University Hospital, Orebro, Sweden
Locations (1):
- Dept. of Orthopedic Surgery and Anesthesia and Intensive Care, Örebro, Sweden

REFERENCES:
- [Derived] Essving P, Axelsson K, Kjellberg J, Wallgren O, Gupta A, Lundin A. Reduced hospital stay, morphine consumption, and pain intensity with local infiltration analgesia after unicompartmental knee arthroplasty. Acta Orthop. 2009 Apr;80(2):213-9. doi: 10.3109/17453670902930008. PMID 19404806